CLINICAL TRIAL: NCT00003627
Title: Phase III Randomized Study of Radiotherapy With or Without Cisplatin and Fluorouracil for Locally Advanced, Nonresectable Squamous Cell Cancer of the Oropharynx or Hypopharynx
Brief Title: Radiation Therapy With or Without Combination Chemotherapy in Treating Patients With Advanced Cancer of the Oropharynx or Hypopharynx
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: UNICANCER (Other)
Responsible Party: Sponsor
Allocation: Randomized | Purpose: Treatment
Other Study IDs: CDR0000066710; FRE-FNCLCC-96003; EU-98027
Record Dates: First submitted 1999-11-01; First posted 2003-04-30 (Estimated); Last update posted 2021-02-21 (Actual); Status verified 2021-02

CONDITIONS: Head and Neck Cancer
Keywords: stage III squamous cell carcinoma of the oropharynx; stage IV squamous cell carcinoma of the oropharynx; stage III squamous cell carcinoma of the hypopharynx; stage IV squamous cell carcinoma of the hypopharynx
MeSH Terms: conditions — Head and Neck Neoplasms; Squamous Cell Carcinoma of Head and Neck | interventions — Cisplatin; Fluorouracil; Radiotherapy

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Drug: cisplatin
Drug: fluorouracil
Radiation: radiation therapy

SUMMARY:
RATIONALE: Radiation therapy uses high-energy x-rays to damage tumor cells. Drugs used in chemotherapy use different ways to stop tumor cells from dividing so they stop growing or die. Combining chemotherapy with radiation therapy may kill more tumor cells and allow doctors to preserve the part of the body where the cancer started. It is not yet known whether radiation therapy with combination chemotherapy is more effective than radiation therapy alone in treating cancer of the oropharynx or hypopharynx that cannot be surgically removed.

PURPOSE: Randomized phase III trial to compare the effectiveness of radiation therapy plus cisplatin and fluorouracil with radiation therapy alone in treating patients who have advanced cancer of the oropharynx or hypopharynx that cannot be surgically removed.

DETAILED DESCRIPTION:
OBJECTIVES:

* Compare the overall survival and survival without relapse for 1, 3, and 5 years of patients with squamous cell cancer of the oropharynx or hypopharynx after treatment with twice a day radiotherapy with or without cisplatin and fluorouracil.
* Compare the presence of distant metastases at 1, 3, and 5 years in these patients after these treatments.
* Compare the local control and duration of control in these patients after these treatments.
* Compare the clinical changes and histological changes at 6 months in these patients after these treatments.
* Determine the rate of complete response in these patients after these treatments.
* Determine the early and late toxic effects of these regimens in these patients.
* Determine the quality of life of these patients.
* Determine the pharmacokinetics of fluorouracil and tolerability of this regimen in these patients.

OUTLINE: This is a randomized, multicenter study. Patients are stratified according to center and primary site of disease (oropharynx vs hypopharynx)

Patients are randomized to one of two treatment arms.

* Arm I: Patients undergo radiotherapy twice a day, 6 hours apart, 5 days a week, for 7 weeks.
* Arm II: Patients undergo radiotherapy as in arm I, plus concurrent chemotherapy consisting of cisplatin IV on day 1 and fluorouracil by continuous infusion over 24 hours on days 1-5. Courses are repeated every 3 weeks for 3 courses.

Patients are followed every month for 1 year, every 2-3 months for 2 years, then every 6 months for at least 2 years.

PROJECTED ACCRUAL: A total of 160 patients (80/arm) will be accrued for this study within 4.5 years.

ELIGIBILITY:
DISEASE CHARACTERISTICS:

* Histologically proven squamous cell cancer of the oropharynx or hypopharynx

  * T4 and nonresectable OR
  * T3 extended to oropharynx or hypopharynx and nonresectable
  * N0-3 (stage III or IV)
* No distant metastases

PATIENT CHARACTERISTICS:

Age:

* 18 to 70

Performance status:

* Karnofsky 70-100%

Life expectancy:

* Greater than 3 months

Hematopoietic:

* Neutrophil count at least 2000/mm^3
* Platelet count at least 100,000/mm^3

Hepatic:

* Bilirubin no greater than 1.25 times upper limit of normal (ULN)
* Transaminases no greater than 2.5 times ULN

Renal:

* Creatinine no greater than 1.25 times ULN

Cardiovascular:

* No severe cardiac disease

Other:

* No prior malignancy except basal cell skin cancer
* No uncontrolled infection

PRIOR CONCURRENT THERAPY:

Biologic therapy:

* Not specified

Chemotherapy:

* No prior chemotherapy
* No concurrent antineoplastic therapy

Endocrine therapy:

* Not specified

Radiotherapy:

* No prior radiotherapy

Surgery:

* No prior surgery (except biopsy or adenectomy)

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 160 (Estimated)
Dates: Start 1998-10 (Actual); Primary Completion 2005-12 (Actual); Study Completion 2011-01 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Rene-Jean Bensadoun, MD, Study Chair — Centre Antoine Lacassagne
Locations (11):
- France (11):
  - Centre Oscar Lambret, Lille
  - Institut J. Paoli and I. Calmettes, Marseille
  - CHU de la Timone, Marseille
  - Centre Regional de Lutte Contre le Cancer - Centre Val d'Aurelle, Montpellier
  - CRLCC Nantes - Atlantique, Nantes-Saint Herblain
  - Centre Antoine Lacassagne, Nice
  - Institut Jean Godinot, Reims
  - Centre Henri Becquerel, Rouen
  - Centre Rene Huguenin, Saint-Cloud
  - Centre Hospitalier Universitaire Bretonneau de Tours, Tours
  - Centre Alexis Vautrin, Vandœuvre-lès-Nancy

REFERENCES:
- [Result] Bensadoun RJ, Benezery K, Dassonville O, Magne N, Poissonnet G, Ramaioli A, Lemanski C, Bourdin S, Tortochaux J, Peyrade F, Marcy PY, Chamorey E, Vallicioni J, Seng H, Alzieu C, Gery B, Chauvel P, Schneider M, Santini J, Demard F, Calais G. French multicenter phase III randomized study testing concurrent twice-a-day radiotherapy and cisplatin/5-fluorouracil chemotherapy (BiRCF) in unresectable pharyngeal carcinoma: Results at 2 years (FNCLCC-GORTEC). Int J Radiat Oncol Biol Phys. 2006 Mar 15;64(4):983-94. doi: 10.1016/j.ijrobp.2005.09.041. Epub 2006 Jan 10. PMID 16376489